CLINICAL TRIAL: NCT01915446
Title: Kidney and Intestinal Markers for Early Detection of Organ Injury After Endovascular Aortic Repair - The KISMED Study
Brief Title: Kidney and Intestinal Markers for Early Detection of Organ Injury After Endovascular Aortic Repair
Acronym: KISMED
Status: Completed | Type: Observational
Sponsor: University Hospital Regensburg (Other)
Responsible Party: Principal Investigator, Professor Hans-Jürgen Schlitt, Prof. Dr. Hans J. Schlitt, University Hospital Regensburg
Other Study IDs: KISMED-001
Record Dates: First submitted 2013-07-31; First posted 2013-08-05 (Estimated); Last update posted 2014-12-18 (Estimated); Status verified 2014-12

CONDITIONS: Ischemia; Fatty Acid-Binding Proteins; Mesenteric Vascular Disease; Acute Kidney Injury
Keywords: EVAR; endovascular aortic repair; acute kidney failure; mesenteric ischemia
MeSH Terms: conditions — Ischemia; Acute Kidney Injury; Mesenteric Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma Urine
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to investigate the predictive value of novel biomarkers and contrast-enhanced ultrasonography for early detection of abdominal end-organ (kidney and intestinum) hypoperfusion and ischemia in patients undergoing endovascular aortic repair (EVAR) for aortic aneurysm or dissection. In this context, patients will be monitored for renal biomarkers (TIMP-2, IGFBP7) and intestinal biomarkers (plasmatic intestinal fatty acid binding protein (i-FABP)) and local tissue perfusion will be assessed using contrast-enhanced ultrasonography (CEUS).

The ultimate goal of this study is an early identification of patients developing one or both of these complications, which may facilitate a timely intervention to improve outcome.

ELIGIBILITY:
Inclusion Criteria:

* Existence of an aortic aneurysm with need of repair as indicated by the treating vascular surgeon
* Aortic stenting involving the origin of both mesenteric (i.e. superior and inferior mesenteric arteries) and kidney arteries
* Central line is present to perform repeated blood collections
* Written informed consent is obtained.

Exclusion Criteria:

* Pre-existing severe liver or kidney injury (defined as spontaneous international normalized ratio (INR) >2 or creatinine >2 mg/dl or renal-replacement therapy in the pre-operative course.)
* Known allergy to ultrasound contrast media (exclusion for the CEUS but not for marker evaluation)
* Anemia with hemoglobin concentration < 7g/dl
* Patients < 18 years of age
* Patients not able to give written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing endovascular aortic repair in a University hospital
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2013-07; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Level of biomarkers of abdominal organ injury (plasmatic i-FABP, TIMP-2, IGFBP7) | 48hours post surgery
  The primary objective of this study is to evaluate the early post-operative course of kidney and intestinal biomarkers in patients following EVAR and their value for prediction of development of acute kidney injury or acute mesenteric ischemia.

SECONDARY OUTCOMES:
Local tissue perfusion and microcirculation as quantified by CEUS | 48 hours post surgery
Incidence of acute kidney injury (AKI) | first 48 hours post surgery
  Incidence of AKI within the first 48 hours as based on current KDIGO/AKIN recommendation (Kidney Disease Improving Global Outcomes - Clinical Practice Guideline for Acute Kidney Injury)
Localization and incidence of intestinal ischemia | first 48 hours post surgery

OTHER OUTCOMES:
Other parameters of postoperative course | in-hospital stay, follow up to 90 days
  * Course of established laboratory markers of hypoperfusion (lactate, creatinine kinase, interleukin 6, C-reactive protein,hemoglobin, central venous oxygen saturation)
  * Standard markers of renal function: serum creatinine (sCr), urine output and estimated glomerular filtration rate (eGFR)
  * Standard Doppler Ultrasound of the kidney vessels and superior mesenteric artery
  * Assessment of hemodynamics (cumulative dose of inotropic support intraoperatively, at 24h and 48h, cumulative fluid balance at 24h, 48h) or pulmonary failure (Horowitz Index)
  * Frequency and localization of other ischemic conditions, such as limb ischemia and cerebral ischemia
  * Identification of an "immunological pattern" indicating intestinal ischemia or kidney failure
  * Severity of illness score SAPS II
  * Need of renal replacement therapy (RRT) in postoperative course (days)
  * Creatinin level and RRT at discharge
  * Length of ICU stay and length of hospital stay - 28- days and 90-days mortality

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Regensburg, Regensburg, Bavaria, Germany

REFERENCES:
- [Derived] Gocze I, Ehehalt K, Zeman F, Riquelme P, Pfister K, Graf BM, Bein T, Geissler EK, Kasprzak P, Schlitt HJ, Kellum JA, Hutchinson JA, Eggenhofer E, Renner P. Postoperative cellular stress in the kidney is associated with an early systemic gammadelta T-cell immune cell response. Crit Care. 2018 Jul 4;22(1):168. doi: 10.1186/s13054-018-2094-x. PMID 29973233